CLINICAL TRIAL: NCT05799820
Title: An Open-label, Multicenter Phase II Study of QL1706 Monotherapy or in Combination With Bevacizumab and XELOX as First-line Treatment of Unresectable Advanced or Metastatic CRC
Brief Title: QL1706 Monotherapy or in Combination With Bevacizumab and XELOX as First-line Treatment of Unresectable Advanced or Metastatic CRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-208
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706 (Experimental)
  Interventions: Drug: QL1706
- QL1706 in combination with bevacizumab and XELOX (Experimental)
  Interventions: Drug: QL1706; Drug: Bevacizumab; Drug: Oxaliplatin injection; Drug: Capecitabine

INTERVENTIONS:
Drug: QL1706 — 5 mg/kg administered as IV infusion on Day 1 of each 21-day cycle
Drug: Bevacizumab — 7.5 mg/kg administered as IV infusion on Day 1 of each 21-day cycle
  Arms: QL1706 in combination with bevacizumab and XELOX
Drug: Oxaliplatin injection — 130mg/m2 administered as IV infusion on Day 1 of each 21-day cycle
  Arms: QL1706 in combination with bevacizumab and XELOX
Drug: Capecitabine — 1000 mg/m2 orally twice daily for 14 days continuous dosing followed by a 7-day break of each 21-day cycle
  Arms: QL1706 in combination with bevacizumab and XELOX

SUMMARY:
This is an open-label, muticenter phase II study to evaluate the efficacy and safety of QL1706 monotherapy or in combination with bevacizumab and XELOX as first-line treatment of unresectable advanced or metastatic CRC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects participate voluntarily and sign informed consent.
* 2. Age ≥ 18 and ≤ 80 years old, male or female.
* 3. Histologically confirmed unresectable locally advanced or metastatic adenocarcinoma of the colon or rectum.
* 4. At least 1 measurable target lesion according to Response Evaluation in Solid Tumors (RECIST 1.1).

Exclusion Criteria:

* 1. Diagnosed additional maliganancy within 5 years with the expection of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin,curatively resected in situ cervival or non-muscle invasive bladder cancers.
* 2. Presence of brain metastases (asymptomatic brain metastases or symptomatic brain metastases who are stable at least 4 weeks, were allowed to be enrolled).
* 3. Has active autoimmune disease that has required systemic treatment in past 2 years.
* 4. Significant cardiovascular disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years
  ORR was assessed by investigators per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to approximately 2 years
  DCR was assessed by investigators per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Duration of Response (DOR) | Up to approximately 2 years
  DOR was assessed by investigators per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Progression-free Survival (PFS) | Up to approximately 2 years
  PFS was assessed by investigators per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Overall Survival (OS) | Up to approximately 2 years
  OS was defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No